CLINICAL TRIAL: NCT04862533
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Beta-alanine and Pelvic Floor Muscle Training on Urinary Incontinence After Radical Prostatectomy (BELA)
Brief Title: Effect of Beta-alanine and Pelvic Floor Muscle Training on Urinary Incontinence After Radical Prostatectomy (BELA)
Acronym: BELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Vladimir Student, M.D., Ph.D., Director of the study, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BELA2020; URIRAPRO(2020) (Other: University Hospital Olomouc)
Record Dates: First submitted 2021-04-19; First posted 2021-04-28 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Urinary Incontinence; Beta-Alanine; Pelvic Floor Muscle Training; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — beta-Alanine; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine + PFMT (Experimental): Participants will ingest an active supplement containing beta-alanine for a period of maximum 6 months. During the whole period, participants will take part in a structured program of PMFT. After first month, the participants will undergo radical prostatectomy.
  Interventions: Drug: Beta-Alanine; Procedure: Pelvic floor muscle training (PFMT)
- Placebo + PFMT (Experimental): Participants will ingest a placebo supplement containing no beta-alanine for a period of maximum 6 months. During the whole period, participants will take part in a structured program of PMFT. After first month, the participants will undergo radical prostatectomy.
  Interventions: Drug: Placebo; Procedure: Pelvic floor muscle training (PFMT)

INTERVENTIONS:
Drug: Beta-Alanine — Participants will receive 1150mg of beta-alanine three times a day
  Other Names: Intervention group
  Arms: Beta-alanine + PFMT
Drug: Placebo — Participants will receive matching placebo three times a day
  Other Names: Control group
  Arms: Placebo + PFMT
Procedure: Pelvic floor muscle training (PFMT) — Participants in both groups will undergo PFMT training program

SUMMARY:
The purpose of this study is to evaluate the effectiveness of beta-alanine in combination with pelvic floor muscle training (PFMT) compared to PFMT plus placebo in men undergoing radical prostatectomy.

DETAILED DESCRIPTION:
This study will assess efficacy of beta-alanine in combination with PFMT for the treatment of participants with urinary incontinence after radical prostatectomy. B-alanine is a component of L-carnosine (with L-histidine), which is needed for its synthesis. Βeta-alanine, thanks to its bioavailability) is a commonly used supplement that can improve exercise performance by increasing the amount of carnosine in striated muscle tissues. Supplementation of beta-alanine in elderly patients has resulted in an increase in physical activity, less fatigue and overall increase in L-carnosine concentration in muscles. PFMT utilization is considered a strong predictor of early return of urinary continence after radical prostatectomy (RP). We hypothesize, that combination of PFMT with beta-alanine could result in improved urinary continence after RP. The intervention will start 30 days before the surgery and will continue until primary outcome is met. Beta-alanine/placebo will be given daily. Efficacy, pharmacokinetics, biomarkers, tissue histology, participants reported outcomes and safety will be assessed. The total duration of study will be approximately 6 months.

ELIGIBILITY:
* Inclusion Criteria:

  * Age 40-80 years
  * Able to give informed consent
  * Histologically proven prostate cancer
  * BMI <35
  * No other cancer treatment
  * Continent
  * Good physical and mental activity
  * On normal diet
  * Scheduled for radical prostatectomy (open or robotic)
* Exclusion Criteria:

  * Other malignant cancer (except for benign skin cancer)
  * Age > 80 years
  * Diabetes mellitus (any type)
  * Chronic bowel inflammatory disease
  * Urinary incontinence
  * Impaired mental activity
  * Previous radiotherapy of hormonal therapy
  * Vegetarian/vegan/on macrobiotic diet

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Time to Continence (days) | up to 6 months
  Continence is defined by number of pads used and measured by one hour pad test. Number of pads use will be determined according to EPIC-SF questionnaire

SECONDARY OUTCOMES:
Assessment of physical activity of participants | up to 6 months
  To assess physical activity of the participants using Physical activity level (PAL), the number of participants having recommended PAL (PAL 1.75: a weekly average PAL of ≥1.75) < 1.4 = extremely inactive, > 2.4 = extremely active
Number of participants with laboratory abnormalities as measure of safety | up to 6 months
  Number of participants with laboratory abnormalities (hematology, serum chemistry and liver function test) will be determined
Number of participants with adverse events | up to 6 months
  Incidence of adverse events in the combined beta-alanine and PFMT compared to PFMT and placebo treatment. Surgical complications will be evaluated according to Clavien-Dindo classification
Assessment of quality of life (QoL) change in both groups of participants | up to 6 months
  During the study period, participants will be asked to fill in clinical validated EuroQuol-5dimensions-5levels (EQ-5D-5L) questionnaire 0 = the worst to 100 = the best QoL outcome
Muscle carnosine concentration | at week 4 (surgery)
  Integrity and architecture of muscle tissue will be assessed in 4 µm thick sections of formalin-fixed, paraffin-embedded, hematoxylin-eosin stained tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Student, MD, PhD, Principal Investigator — Dpt. of Urology, University hospital Olomouc
Locations (1):
- University hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No